CLINICAL TRIAL: NCT00530829
Title: Clinical Effectiveness and Preventive Impact of Home Zinc Treatment for Acute Diarrhea in Children: A Cluster-randomized Field Trial in Rural Western Kenya
Brief Title: Impact of Home Zinc Treatment for Acute Diarrhea in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kenya Medical Research Institute (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Daniel Feikin, Medical epidemiologist, CDC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCPDCID-4678
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Diarrhea
Keywords: diarrhea; zinc; oral rehydration therapy
MeSH Terms: conditions — Diarrhea | interventions — Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Mothers recieve a blister pack of zinc tablets in home every two months for use when child in home under 5 years has diarrhea. ORS satchets also given. Instructions on when and how to use zinc and ORS and when to take child in clinic are given by community health worker. Zinc will also be given in clinic if child visits clinic with diarrhea and has not yet started zinc at home.
  Interventions: Drug: zinc
- 2 (Active Comparator): Mothers recieve ORS satchets at home every two months for use when child in home under 5 years has diarrhea. Instructions on when and how to use ORS and when to take child in clinic are given by community health worker. Zinc will be given in clinic if child visits clinic with diarrhea.
  Interventions: Drug: zinc

INTERVENTIONS:
Drug: zinc — 10 day blister pack of 20 mg zinc disperable tablets, 1 tablet qd for children 6 months to 4 years, 1/2 tablet qd for children 2-5 months

SUMMARY:
Background. Zinc deficiency is common in Africa. It has been shown in Asia that zinc as treatment for diarrhea can shorten the course of episodes of diarrhea, as well as prevent future episodes. The use of zinc at home to treat diarrhea in an African setting, where malaria, HIV and malnutrition are common, has not been well-studied.

Objective. To evaluate if zinc treatment for diarrhea given at home in Kenyan children will decrease the community prevalence of diarrhea more than zinc given only in the clinic Work planned. We propose to do a community-randomized intervention study of 10 days of dispersible zinc tablets given in the home, in addition to ORS, to treat diarrhea in children under-5 years of age living in a rural part of Bondo District. The comparison group will be children who receive zinc and ORS in the clinic only. The primary outcome will be a comparison of the prevalence of diarrhea in home zinc versus nonhome zinc villages. Secondary outcomes will be the incidence of repeat episodes of diarrhea, the duration of diarrheal illness, the prevalence of acute respiratory infection, and the effect of malaria infection on treatment with zinc. Thirty-three villages (approximately 1300 children) will be enrolled and children will be followed for 1 year.

Significance of results. If this study shows zinc given at home to be effective, this might be considered by the Kenyan MOH as an essential component of the treatment of diarrhea in children at the community level.

ELIGIBILITY:
Inclusion Criteria:

* All children 2 to 59 months of age in households within 33 selected villages

Exclusion Criteria:

* Children under 2 months of age will not be eligible for enrollment, until they reach 2 months of age as the role of zinc has not been well-studied in neonates. Children of parents who do not give written informed consent for their participation will not be enrolled.

Ages: 2 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To assess if access to zinc treatment for diarrhea in the home in addition to zinc treatment of diarrhea in the clinic leads to a greater reduction in the prevalence of diarrhea than giving zinc for treatment of diarrhea in the clinic only | One year

SECONDARY OUTCOMES:
To assess if access to zinc treatment for diarrhea in the home in addition to zinc treatment of diarrhea in the clinic decreases the likelihood of recurrent diarrhea episodes, acute respiratory infections, and antimicrobial use | one year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Feikin, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

REFERENCES:
- [Derived] Feikin DR, Bigogo G, Audi A, Pals SL, Aol G, Mbakaya C, Williamson J, Breiman RF, Larson CP. Village-randomized clinical trial of home distribution of zinc for treatment of childhood diarrhea in rural Western kenya. PLoS One. 2014 May 16;9(5):e94436. doi: 10.1371/journal.pone.0094436. eCollection 2014. PMID 24835009
- See also: Document WHO/FCH/CAH/04.7 — http://www.who.int